CLINICAL TRIAL: NCT00760890
Title: Iron and the Breast-Fed Infant: Iron Status and Two Regimens of Iron Supplementation
Acronym: BFe01B1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health (NIH) (NIH)
Responsible Party: Ekhard E. Ziegler, M.D., University of Iowa
Organization: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD040315 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Iron Deficiency
Keywords: Iron, breastfed infant
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

ARMS (3):
- A (Experimental): Medicinal Iron
  Interventions: Dietary Supplement: Fer-In-Sol (ferrous sulfate)
- B (Experimental): Iron fortified wet pack cereal
  Interventions: Dietary Supplement: Iron fortified cereal
- C (No Intervention): Control

INTERVENTIONS:
Dietary Supplement: Fer-In-Sol (ferrous sulfate) — 7.5 mg/day in the form of 0.3 ml once each day
  Arms: A
Dietary Supplement: Iron fortified cereal — 1 jar each day of one of three wet pack cereals manufactured by the Gerber Company: Each jar provided 7 mg of ferrous sulfate.
  Arms: B

SUMMARY:
Normal breastfed infants can develop iron deficiency by 6 months of age. This trial tested the hypothesis that regular provision of a source of iron beginning at 4 months of age improves iron status and could prevent iron deficiency. This was a prospective randomized trial involving breastfed infants. To be eligible, infants had to be predominantly breastfed (<200 ml/day of formula) at 4 months of age. At 4 months infants were randomly assigned to one of two interventions or to control. The interventions consisted in the daily administration of medicinal iron in a dose of 7.5 mg (Medicinal Iron Group) or in the daily feeding of one jar of an iron-fortified cereal providing 7 mg of iron each day (Cereal Group). The control group received complementary foods chosen by he parents but no source of iron provided by the investigators. The interventions took place from 4 to 9 months. All infants were subsequently followed to 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Predominantly breastfed (at 4 months) term infants

Exclusion Criteria:

* Not predominantly breastfed at 4 months
* Premature infants

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2001-06; Primary Completion 2005-06 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Iron status | 3 times during the intervention

SECONDARY OUTCOMES:
Growth | At the end of intervention
Tolerance (gastrointestinal) | During intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ekhard E Ziegler, M.D., Principal Investigator — University of Iowa
Locations (1):
- Fomon Infant Nutrition Unit, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Ziegler EE, Nelson SE, Jeter JM. Iron status of breastfed infants is improved equally by medicinal iron and iron-fortified cereal. Am J Clin Nutr. 2009 Jul;90(1):76-87. doi: 10.3945/ajcn.2008.27350. Epub 2009 May 20. PMID 19458014